CLINICAL TRIAL: NCT01374490
Title: A Phase 3, Multicenter, Open-Label Evaluation of the Safety and Tolerability of Crofelemer in HIV-Positive Subjects With Diarrhea
Brief Title: Safety and Tolerability of Crofelemer for HIV-Associated Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFHD3092
Record Dates: First submitted 2011-06-13; First posted 2011-06-16 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: HIV Enteropathy; Diarrhea With HIV
Keywords: HIV +; HIV positive; HIV associated diarrhea; AIDS; Diarrhea
MeSH Terms: conditions — HIV Enteropathy; HIV Seropositivity; Acquired Immunodeficiency Syndrome; Diarrhea | interventions — crofelemer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Crofelemer (Experimental)
  Interventions: Drug: Crofelemer

INTERVENTIONS:
Drug: Crofelemer — Crofelemer will be administered orally as 1 tablet(125 mg)BID for a total daily dose of 250mg crofelemer.

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of crofelemer 125 mg twice a day, taken orally, over 48 weeks of therapy in human immunodeficiency virus-positive (HIV+) subjects with diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* History of HIV-1 infection
* On an antiretroviral therapeutic regimen for treatment of HIV-1 disease and associated conditions (including prophylactic antibiotics for Pneumocystis jirovecii or infection) for at least 4 weeks prior to screening
* Self-reported presence of diarrhea necessitating ADM use for at least 4 weeks

Exclusion Criteria:

* CD4 counts < 100 cells/mm3
* Oral temperature greater than 38.0° C, or unintentional weight loss of 5.0 kg or greater during the prior 2 months
* Bright red blood per rectum judged not to be of an anal (e.g., hemorrhoid, fissure) origin
* Immediate need for GI surgery or intervention for active GI bleeding, pancreatitis, peritonitis, intestinal obstruction, or intra-abdominal abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Beverly Hills, California
  - Los Angeles, California
  - San Diego, California
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Wilton Manors, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Detroit, Michigan
  - Santa Fe, New Mexico
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crofelemer
Started | 250
Completed | 190
Not Completed | 60

BASELINE CHARACTERISTICS:
Arm/Group | Crofelemer
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 211

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs).
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer
Number analyzed (Participants) | 250
Participants
  Any TEAE | 189
  Any SAEs | 20

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Crofelemer
Serious Adverse Events (participants affected / at risk) | 20/250
Other Adverse Events (participants affected / at risk) | 107/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crofelemer (N=250)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
ABSCESS LIMB (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 4
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 1
GASTROENTERITIS CRYPTOSPORIDIAL (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CONVULSION (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
HYPERTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crofelemer (N=250)
Constipation (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 14
Upper respiratory tract infection (Infections and infestations) | 42
Parasitic infection intestinal (Infections and infestations) | 31
Giardiasis (Infections and infestations) | 20
Bronchitis (Infections and infestations) | 15
Blastocystis infection (Infections and infestations) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details